CLINICAL TRIAL: NCT03829137
Title: The Clinical Effects of Laser Acupuncture Therapy for OAB Women: a Randomized Controlled Trial.
Brief Title: The Clinical Effects of Laser Acupuncture Therapy for OAB Women.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201801679A3
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum laser acupuncture (Experimental): Verum laser acupuncture：Low level laser therapy stimulates 7 acupuncture points on both sides of the body .
  Interventions: Device: Verum laser acupuncture
- Sham laser acupuncture (Sham Comparator): sham laser acupuncture (no laser output)
  Interventions: Device: Sham laser acupuncture

INTERVENTIONS:
Device: Verum laser acupuncture — The patients lay in the supine position before treatment and the gallium aluminum arsenide LaserPan (RJ-Laser, Reimers & Janssen GmbH, Waldkirch, Germany) will be applied to each selected acupoints for 3 weeks, total of 9 sessions.
  Arms: Verum laser acupuncture
Device: Sham laser acupuncture — The acupuncture points and procedure of the control group are identical to the experimental group but there are no laser beam energy.
  Arms: Sham laser acupuncture

SUMMARY:
Overactive bladder (OAB) is a syndrome causes urgency, with or without urgent incontinence, daytime frequency and nocturia. Urgency incontinence is more common in older women and may be associated with comorbid conditions that occur with age. The standard OAB medical treatments may induced several intolerable side effects including dry mouth, constipation, and so on, therefore alternative therapies are often considered. Acupuncture had been proved effective to OAB treatment, however, this invasive procedure also cause pain and hematoma. Laser acupuncture has minimal side effects comparing to conventional acupuncture, but its effects against OAB had never been examined. Experiments with laser acupuncture are expected to be another way to relieve OAB symptoms.

DETAILED DESCRIPTION:
The subjects are treated with 7 acupoints which are localized according to WHO standardized acupressure point location guideline. The patients lay in the supine position before treatment and the gallium aluminum arsenide LaserPan (RJ-Laser, Reimers & Janssen GmbH, Waldkirch, Germany) will be applied to each selected acupoints mentioned above. The experimental group (verum laser acupuncture) and control group (sham laser acupuncture) will receive laser acupuncture 3 times per week for 3 weeks, total of 9 sessions, based on clinical experience (Treatment could be extended if necessary). The basic patient data will be recorded at baseline and adverse effect will also be recorded during the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Women are older than 18 years old.
2. Participant is willing to sign the consent.
3. Women havea moderate OAB symptoms.
4. Total scores of OABSS > 6 points and the 3rd question of OABSS > 2 points.
5. Not using anticholinergic drugs for more than three weeks.

Exclusion Criteria:

1. Patients with lower urinary tract infection.
2. Patients who cannot complete the questionnaire.
3. Patients who use Botox to inject bladder and pelvic floor muscles within one year.
4. Pregnant patients.
5. Patients who continue to have electrical stimulation and acupuncture in the legs, waist and pelvis.
6. Patients with vaginal bleeding.
7. Other herbal and folklore therapies are being used to improve patients with overactive bladder.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-04-05 (Estimated); Study Completion 2022-04-05 (Estimated)

PRIMARY OUTCOMES:
OAB symptom score (OABSS) | 3 weeks
  This is a four symptoms questionnaire to quantify OAB symptoms.

SECONDARY OUTCOMES:
The Urogenital Distress Inventory (UDI-6) | 3 weeks
  This evaluation scale assesses symptom distress.

OTHER OUTCOMES:
Incontinence Impact Questionnaire (IIQ-7) | 3 weeks
  This evaluation scale assesses the impact on daily life of urinary incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Ning Chang, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No